CLINICAL TRIAL: NCT00811174
Title: Clinical Study to Evaluate the Efficacy, Safety and Kinetics of Octagam 10% for Replacement Therapy in Primary Immunodeficiency Diseases
Brief Title: Efficacy, Safety and Kinetics Study of Octagam 10% in Primary Immunodeficiency Diseases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to limited data available, efficacy, and PK analyses were not performed.
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAM10-03
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Immunologic Deficiency Syndromes
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Octagam 10% (Experimental)
  Interventions: Drug: Octagam 10%

INTERVENTIONS:
Drug: Octagam 10% — 300-600 mg/kg every 21 (+/- 3 days) to 28 days (+/- 3 days)

SUMMARY:
Octagam is a human normal immunoglobulin (IGIV) solution for intravenous administration. Octagam 5% is currently registered in more than 60 countries. This study will evaluate the efficacy, safety and the kinetics of Octagam 10% for replacement therapy in primary immunodeficiency diseases.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the safety of Octagam 10% in replacement therapy in PID and to compare the pharmacokinetic profile of Octagam 10% with that of the previously used Octagam 5%.

The secondary objective is to investigate the efficacy of Octagam 10% in replacement therapy in PID by monitoring the rate of occurence of serious bacterial infections, the rate of other infections, the trough (pre-next-dose) levels of total serum IgG and IgG subclasses (IgG1, IgG2, IgG3 and IgG4), the trough (pre-next-dose) levels of selected antigen specific antibodies, the use of antibiotics, the rate of absence from school/ work, and the number of days in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary immunodeficiency (acc. WHO)
* Previous treatment with commercial Octagam 5% every 3-4 weeks for at least 6 infusions intervals
* Documented IgG trough levels of the two previous infusions before enrollment with a value of at least 5.5 g/L for both

Exclusion Criteria:

* Acute infection requiring intravenous antibiotic treatment within two weeks before screening
* Exposure to blood or any blood product or derivative other than commercially available Octagam 5%, within the past 3 months
* History of hypersensitivity to blood or plasma derived products
* Requirement of any routine premedication for IGIV treatment
* History of congenital impairment of pulmonary function
* Severe liver function impairment
* Severe renal function impairment or predisposition for acute renal failure
* History of autoimmune haemolytic anaemia
* History of diabetes mellitus
* Congestive heart failure NYHA III or IV
* Non-controlled arterial hypertension
* History of DVT or thrombotic complications with IGIV treatment
* Known infection with HIV, HCV or HBV
* Treatment with steroids, immunosuppressive or immunomodulatory drugs
* Planned vaccination during study period
* Pregnant or nursing woman

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Dr., Study Director — Octapharma
Locations (1):
- Contact Barbara Pyringer at Octapharma/ Vienna/ Austria for information, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients previously treated with commercial Octagam 5% were to be enrolled in the study on the basis of the in- and exclusion criteria defined in the study protocol. Patients were to be enrolled only after written informed consent by the patient had been obtained.
Groups:
- Octagam 10%: Octagam 10% : 300-600 mg/kg every 21 (+/- 3 days) to 28 days (+/- 3 days)
Period: Overall Study
Arm/Group | Octagam 10%
Started | 5
Completed | 2
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Sponsors Decision | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated prematurely. Owing to the limited data available (only 5 patients enrolled, of whom 2 completed the study and 3 ended treatment prematurely), efficacy and PK analyses were not performed. The safety analysis did not yield any unexpected results suggestive of a change in the risk-benefit evaluation of Octagam 10%.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Occurrence of Adverse Events
Time Frame: During infusion or within 72 hours after end of infusion
Measure: Number; unit: participants
Arm/Group | Octagam 10%
Number analyzed (Participants) | 5
participants | 4

2. Primary Outcome: Pharmacokinetics of Serum Total IgG and IgG Subclasses (IgG1, IgG2, IgG3 and IgG4) and Pharmacokinetics of Specific Antibodies Against Defined Infectious Agents Comparing Octagam 5% Treatment With Octagam 10% Treatment
Description: Pharmacokinetics of serum total IgG and IgG subclasses (IgG1, IgG2, IgG3 and IgG4) and pharmacokinetics of specific antibodies against defined infectious agents comparing Octagam 5% treatment with Octagam 10% treatment
Time Frame: after 6 months of treatment
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

3. Secondary Outcome: Vital Signs
Time Frame: during each treatment
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

4. Secondary Outcome: Laboratory Parameters (Hematology, Clinical Chemistry, Direct Coombs Test and Urin Analysis)
Time Frame: at each treatment date (every three to four weeks)
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

5. Secondary Outcome: Assessment of Viral Safety
Time Frame: Every three months
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

6. Secondary Outcome: Pre-next-dose Levels of Serum Total IgG
Time Frame: before each treatment
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

7. Secondary Outcome: Pre-next-dose Levels of IgG Subclasses (IgG1, IgG2, IgG3, IgG4) and Pre-next-dose Levels of Specific Antibodies Against Defined Infectious Agents
Time Frame: before treatement 10 and 13 (of 13 or 17 treatments) and at the end
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

8. Secondary Outcome: Therapeutic Efficacy (Number of Infections, Number of Missed Days at School/ Work, Number of Hospitalisation Days, and Use of Antibiotics)
Time Frame: 12 months
Population: Due to premature termination of the study, data were unavailable and no analysis was done.
Arm/Group | Octagam 10%
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Description: In summary, the assessment of adverse events, laboratory variables and other safety-related observations revealed no reasons for concern about the safety of Octagam 10%.
Arm/Group | Octagam 10%
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octagam 10% (N=5)
surgery for inguinal condyloma (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octagam 10% (N=5)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
upper respirotory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
gastroenteritis (Gastrointestinal disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pharyngolarynngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No